CLINICAL TRIAL: NCT05741021
Title: A Single-arm, Open-label, and Multicenter Phase Ⅱ Study Designed to Evaluate the Efficacy and Safety of Rulonilimab Combined With Chemotherapy in Patients With Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase II Study of Rulonilimab Combined With Chemotherapy in the First-Line Treatment for Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F520-103
Record Dates: First submitted 2023-02-12; First posted 2023-02-23 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Non-small Cell Lung Cancer; NSCLC; PD-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Rulonilimab+Chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F520+Chemotherapy (Experimental): Cohort 1:
  Treatment period (3 weeks/cycle): On the first day of each cycle, F520 (200 mg), pemetrexed and carboplatin were administered sequentially by intravenous infusion (at least 30 min between doses).
  Maintenance period (3 weeks/cycle): On the first day of each cycle, F520 (200 mg) and pemetrexed were administered sequentially by intravenous infusion (at least 30 min between doses).
  Cohort 2:
  Treatment period (3 weeks/cycle): On the first day of each cycle, F520 (200 mg), paclitaxel and carboplatin were administered sequentially by intravenous infusion (at least 30 min between doses).
  Maintenance period (3 weeks/cycle): On the first day of each cycle, F520 (200 mg) was administered sequentially by intravenous infusion (at least 30 min between doses).
  Interventions: Drug: F520; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: F520 — F520 is a recombinant, humanized programmed death receptor-1 (PD-1) monoclonal antibody that binds to PD-1 and prevents binding of PD-1 with programmed death ligands 1 (PD-L1) and 2 (PD-L2).
  Other Names: Rulonilimab
Drug: Pemetrexed — A chemotherapy medication used to treat a number of types of cancer.
Drug: Carboplatin — A chemotherapy medication used to treat a number of types of cancer.
Drug: Paclitaxel — A chemotherapy medication for the treatment of pleural mesothelioma and non-small cell lung cancer (NSCLC).

SUMMARY:
This is a single-arm, open-label, and multicenter phase Ⅱ study designed to evaluate the efficacy and safety of rulonilimab combined with chemotherapy in patients with advanced or metastatic non-small cell lung Cancer (NSCLC). Two cohorts were designed in this study: cohort 1 (non-squamous NSCLC) and cohort 2 (squamous NSCLC). About 84 patients with advanced or metastatic NSCLC plan to be enrolled in about 20 study sites of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years;
2. Understand and voluntarily sign the written informed consent form;
3. Study population:

   Patients with histologically or cytologically confirmed locally advanced (stage IIIB/IIIC) or metastatic (stage IV) NSCLC who cannot receive surgery or radical concurrent chemoradiotherapy, based on the "8th Edition of the TNM Classification for Lung Cancer" issued by the International Association for the Study of Lung Cancer (IASLC); Have not received any prior systemic anti-tumor therapy for advanced/metastatic disease; Subjects who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of stage IIIB, IIIC, IV.

   Without mutation of epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK) or ROS-1; Note: The results of blood tests alone were not accepted;
4. With a life expectancy of more than 3 months;
5. With at least one measurable lesion (extra nodal lesions: long diameter > 10 mm, nodal lesions: long diameter > 15 mm) confirmed by contrast-enhanced CT or MRI according to RECIST v1.1;
6. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1;
7. Vital organ functions meet the following requirements (Reception of granulocyte colony-stimulating factor (G-CSF) or pegylated granulocyte colony-stimulating factor (PEG-G-CSF) or blood transfusion within 14 days prior to laboratory tests is not permitted for prophylactic use):

   Blood routine examination: absolute neutrophil count (ANC) ≥ 1.5×109/L, hemoglobin (HGB) ≥ 90g/L, platelet count (PLT) ≥ 100×109/L; Hepatic function: total bilirubin (TBIL) ≤ 1.5×ULN, and alanine transaminase (ALT) and aspartate amino transferase (AST) ≤ 2.5×ULN for all patients, or AST and ALT levels ≤ 5×ULN for patients with liver metastases; Renal function: serum creatinine (Cr) ≤ 1.5×ULN or clearance of creatinine (CCr) ≥ 60 mL/min (Cr > 1.5×ULN); Coagulation function: international normalized ratio (INR) ≤ 1.5×ULN and Activated partial thromboplastin time (APTT) ≤ 1.5×ULN； Thyroid stimulating hormone (TSH) is within the normal range; If TSH is abnormal, free triiodothyronine (FT3) and free thyroxine (FT4) should be normal or abnormal without clinical significance;
8. Have provided tumor tissue specimens at or after the diagnosis of advanced or metastatic disease (Formalin-fixed, paraffin-embedded (FFPE) tumor tissues that were archived or freshly obtained within 6 months before the first dose; Tissue specimens require PD-L1 expression to be evaluable).

Exclusion Criteria:

1. Cohort 1: Have a histologically confirmed diagnosis of NSCLC with predominant squamous cells; Patients with mixed histology are not allowed if there is small cell component in the specimen; Cohort2: Have a histologically confirmed diagnosis of NSCLC with predominant Non-squamous cells; Mixed tumors will be categorized by the predominant cell type; if small cell carcinoma, neuroendocrine carcinomas and sarcomas elements are present, the subject is ineligible; Patients with mixed histology are allowed if there is squamous component >50% in the specimen.
2. Has active central nervous system (CNS) metastases and/or carcinomatous meningitis in the past or during screening, except for the following cases:

   Subjects with asymptomatic brain metastases (i.e., no neurological symptoms, no requirements for corticosteroids, and no lesion >1.5 cm) may participate but will require regular imaging of the brain as a site of disease; Subjects with adequate treatmen may participate provided they are clinically stable for at least 4 weeks, and his nervous system and other clinical symptoms can return to the baseline level at least 2 weeks before the first dose (Except for residual signs or symptoms related to CNS therapy).
3. Subjects with spinal cord compression not curatively cured by surgery and/or radiotherapy.
4. Had prior treatment with anti-PD-1, or PD-L1, or PD-L2, or CD137, or CTLA-4 antibody or fusion protein or any other antibodies or drugs that specifically target T cell co-stimulatory or checkpoint pathways.
5. Have suffered from interstitial lung disease, non-infectious pneumonia or uncontrolled lung disease in the past 3 years, including but not limited to pulmonary fibrosis, acute lung disease, etc. (Except chemotherapy-induced interstitial lung disease that is currently asymptomatic).
6. Patients with uncontrolled or severe cardiovascular diseases, such as Class II-IV congestive heart failure, unstable angina, myocardial infarction and other cardiovascular diseases assessed by New York Heart Association (NYHA), uncontrolled hypertension (systolic blood pressure ≥ 180mmHg and/or diastolic pressure ≥ 100mmHg), poorly controlled arrhythmia (Including QTc interval male ≥ 450 ms, female ≥ 470 ms) within 6 months before the first dose.
7. Subjects with symptomatic ascites, pericardial effusion or pleural effusion whose clinical status is stable for more than 1 month after receiving treatment (including therapeutic chest X-ray or puncture) can be enrolled.
8. Subjects who are using or have recently used (within 7 days before the first dose of study drug) aspirin therapy, or is unable to interrupt nonsteroidal anti-inflammatory drugs (NSAIDs) during the study. (apply to cohort 1)
9. Is unable or unwilling to take folic acid or vitamin B12 supplementation; Is unable to take corticosteroids; (Apply to cohort 1)
10. Has the following conditions in physical examination and laboratory examination:

    With a known positive history of human immunodeficiency virus (HIV), Has known history of Human Immunodeficiency Virus (HIV) positive or acquired immunodeficiency syndrome (AIDS); Subjects with positive for treponema pallidum (TP) antibody； With active hepatitis, hepatitis B: HBsAg positive and/or HBcAb positive,a nd HBV-DNA level positive or above the ULN; hepatitis C: HCV antibody positive and HCV-RNA level positive or above the ULN;
11. Has a known contraindications or history of hypersensitivity to any component of test drug or to any excipients.
12. Has received organ in the past or autologous stem cell transplantation within 3 months before the first dose.
13. Received radiation therapy to the lung in the past.
14. Has other history of malignancy within the past 3 years, except locally curable cancer (such as radical melanoma, basal or squamous cell carcinoma, in situ cancer of the bladder or cervix).
15. Has received any drugs with anti-cancer indications (including Chinese herbal or patent medicine, immunosuppressants, systemic or topical hormones) for immunosuppression within 14 days before the first dose (Daily dose of systemic corticosteroid equivalent to prednisone >10 mg).
16. Had major surgery (<28 days prior to first dose) or have not recovered from major surgery.
17. Has active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
18. Patients with unexplained fever > 38.5°C during the screening period and before the first dose (judged by the investigator, patients with fever due to tumors can be enrolled).
19. Received any other study therapy (drugs or devices) within 4 weeks prior to first dose.
20. Had a history of substance abuse or alcoholism (<6 months prior to first dose).
21. Have received a live-virus vaccination within 28 days prior to the first dose or plan to receive a live-virus vaccination during the study (Inactivated virus vaccines such as injectable seasonal flu vaccine and COVID-19 vaccine are allowed during the study period).
22. Is pregnant or breastfeeding; Female of childbearing potential or male with a female partner(s) of child-bearing potential is unwillingness to use effective contraception measures during the study or through 6 months after last dose.
23. The investigator believes that it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-10-25 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  ORR (CR+PR) as assessed by the investigator per RECIST v1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years
  OS defined as the time from the date of randomization to the date of death due to any cause.
Progression-free survival (PFS) | up to 2 years
  PFS as assessed by the investigator per RECIST v1.1.
disease control rate (DCR) | up to 2 years
  DCR as assessed by the investigator per RECIST v1.1.
Duration of remission (DOR) | up to 2 years
  DOR as assessed by the investigator per RECIST v1.1.
Time to progression (TTP) | up to 2 years
  TTP as assessed by the investigator per RECIST v1.1.
Incidence and severity of adverse events (AEs) | up to 2 years
  All toxicities or AEs graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), v5.0.
Incidence and severity of serious adverse events (SAEs) | up to 2 years
  All toxicities or AEs graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), v5.0.

OTHER OUTCOMES:
the positive rate of ADA | up to 2 years
  Explore immunogenicity
the positive rate of neutralizing antibodies | up to 2 years
  Explore the positive rate of neutralizing antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No